CLINICAL TRIAL: NCT04978883
Title: Characteristics of Patients With Primary Sjögren's Syndrome Associated Interstitial Lung Disease and Relevant Features of Disease Progression
Brief Title: Interstitial Lung Diseases in Primary Sjogren's Syndrome
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 20181236FSKXJ
Record Dates: First submitted 2021-07-18; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pSS-ILD: diagnosis of pSS-ILD was based on abnormal HRCT and PFTs
  Interventions: Other: No intervention
- pSS non-ILD: pSS patients after exclusion of pSS-ILD and concomitant pulmonary diseases were considered as pSS non-ILD
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Patients with pSS seen in the Division of Rheumatology, the second affiliated hospital of Zhejiang University, School of Medicine (SAHZU) during January 2016 to July 2018, were retrospectively reviewed. Characteristics were analyzed.

DETAILED DESCRIPTION:
Patients with pSS were retrospectively reviewed, and pSS-ILD and pSS non-ILD were identified. Clinical data, laboratory parameters, pulmonary high-resolution CT (HRCT), and pulmonary function tests (PFTs) were collected. pSS-ILD patients were further categorized into subgroups according to HRCT patterns or PFTs.

ELIGIBILITY:
Inclusion Criteria:

* All patients with pSS fulfilled the 2002 revised version of the European criteria proposed by the American-European Consensus Group
* Patient with pSS evaluated with pulmonary HRCT and/or PFTs were included in the pSS-ILD group

Exclusion Criteria:

* patients with hepatitis C infection, past head and neck radiation treatment, sarcoidosis, acquired immunodeficiency syndrome, pre-existing lymphoma, graft-versushost disease, and use of anticholinergic drugs, IgG4-related disease
* Patients with other connective tissue diseases (CTD) or other pulmonary diseases were further excluded, including those with pulmonary arterial hypertension, pulmonary infections, tuberculosis, chronic bronchitis, emphysema, asthma, chronic obstructive pulmonary disease, malignancies, pulmonary lesions related with environmental, occupational or medication exposures, or history of smoking

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eighty-five patients with pSS-ILD were identified, and 85 patients with pSS non-ILD were used for comparison. The average age at disease onset and median disease duration in patients with pSS-ILD were greater when compared with pSS non-ILD patients. There was no difference regarding presenting symptoms at disease onset between pSS-ILD and pSS non-ILD patients.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
observational study, data analysis to identify the risk factors of pSS-ILD | 6 months from baseline
  ILD progressed in 6 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Chen, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University

IPD SHARING:
Plan to Share IPD: No